CLINICAL TRIAL: NCT02579135
Title: Reducing HIV Risk Among Adolescents: Evaluating Project HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laura Widman, Assistant Professor, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 57033; R00HD075654 (NIH)
Record Dates: First submitted 2015-10-10; First posted 2015-10-19 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: HIV; Sexually Transmitted Diseases
Keywords: Condoms; Sexual Abstinence; Sexual Communication
MeSH Terms: conditions — Sexually Transmitted Diseases; Sexual Abstinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project HEART (Experimental): Interactive website with five modules to address safer sex motivation, knowledge, attitudes/norms, self-efficacy, and sexual communication skills. Program takes approximately 30-45 minutes to complete.
  Interventions: Behavioral: Safer Sex
- Control: Project Growing Minds (Other): Attention-matched control website with five modules to address an introduction to mindsets, growth mindsets of intelligence, growth mindsets of self-control, growth mindsets of people, and an integrative summary. Program takes approximately 30-45 minutes to complete.
  Interventions: Behavioral: Growth Mindsets

INTERVENTIONS:
Behavioral: Safer Sex — Interactive web-based intervention with five modules: motivation, knowledge, attitudes/norms, self-efficacy, and sexual communication skills.
  Arms: Project HEART
Behavioral: Growth Mindsets — Interactive web-based intervention with five modules: mindsets introduction, growth mindsets of intelligence, growth mindsets of self-control, growth mindsets of people, and integrative summary.
  Arms: Control: Project Growing Minds

SUMMARY:
This study evaluates an educational web-based intervention designed to increase adolescent girls' motivation and skills to engage in safer sexual behavior (Project HEART: Health Education and Relationship Training). Half of participants will receive Project HEART and half of participants will receive Project Growing Minds, an attention-matched control website focused on growth mindsets of intelligence and self-regulation. The ultimate goal of this work is to help girls reduce their risk of HIV and other sexually transmitted diseases and to avoid unplanned pregnancies.

DETAILED DESCRIPTION:
This study evaluates an educational web-based intervention designed to increase adolescent girls' motivation and skills to engage in safer sexual behavior (Project HEART: Health Education and Relationship Training). Half of participants will receive Project HEART and half of participants will receive Project Growing Minds, an attention-matched control website focused on growth mindsets of intelligence and self-regulation. The ultimate goal of this work is to help girls reduce their risk of HIV and other sexually transmitted diseases and to avoid unplanned pregnancies.

Primary outcomes for this study include 1) acceptability of the program, 2) communication self-efficacy, and 3) communication intentions.

ELIGIBILITY:
Inclusion Criteria:

* 10th grade girl
* Able to read English

Exclusion Criteria:

* None

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 222 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2016-05-04 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Widman, PhD, Principal Investigator — North Carolina State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

REFERENCES:
- [Derived] Widman L, Golin CE, Kamke K, Burnette JL, Prinstein MJ. Sexual Assertiveness Skills and Sexual Decision-Making in Adolescent Girls: Randomized Controlled Trial of an Online Program. Am J Public Health. 2018 Jan;108(1):96-102. doi: 10.2105/AJPH.2017.304106. Epub 2017 Nov 21. PMID 29161072
- [Derived] Widman L, Golin CE, Noar SM, Massey J, Prinstein MJ. ProjectHeartforGirls.com: Development of a Web-Based HIV/STD Prevention Program for Adolescent Girls Emphasizing Sexual Communication Skills. AIDS Educ Prev. 2016 Oct;28(5):365-377. doi: 10.1521/aeap.2016.28.5.365. PMID 27710087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Project HEART | Control: Project Growing Minds
Started | 107 | 115
Completed | 105 | 106
Not Completed | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Project HEART | Control: Project Growing Minds | Total
Number analyzed (Participants) | 107 | 115 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.26 (.48) | 15.22 (.47) | 15.24 (.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 115 | 222
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic | 38 | 45 | 83
  Black/Non-Hispanic | 29 | 25 | 54
  Hispanic | 31 | 34 | 65
  Other/Mixed Race-Ethnicity | 9 | 11 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 107 | 115 | 222

OUTCOME MEASURES:

1. Primary Outcome: 6-item Self-report of Program Acceptability
Description: Program acceptability was assessed through a questionnaire that was adapted from prior acceptability surveys. Specifically, six items were included to assess six aspects of acceptability: (i) an intent to return to the website, (ii) whether one would recommend the program to a friend, (iii) whether one would use information from the program in the future, (iv) how much one liked the program, (v) how much one learned from the program and (vi) how much one felt the program kept their attention. The first three questions were coded with dichotomous response options (yes/no-unsure), whereas the last three items used a four point Likert-type scale ranging from 1=not at all to 4=a lot. For analyses, these last 3 items were dichotomized into 1=a lot and 0=not a lot.
Time Frame: Immediate post-test at completion of intervention
Population: Data on acceptability only analyzed among girls who completed the Project HEART intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Project HEART
Number analyzed (Participants) | 107
Participants
  Would return to site | 84
  Recommend to friend | 94
  Use Information in Future | 101
  Liked program a lot | 60
  Learned a lot | 80
  Program kept attention a lot | 69

2. Primary Outcome: 7-item Self-report of Sexual Communication Self-efficacy
Description: We used the validated Self-Efficacy for HIV Prevention Scale to assess communication self-efficacy. Seven items assessed confidence communicating about sexual topics (e.g., "How sure are you that you could talk to your partner about safer sex?"). Participants responded from 1 for "couldn't do it" to 4 for "very sure." Scores were averaged with higher scores indicating greater confidence in communicating about sex (alpha = 0.82).
Time Frame: Immediate post-test at completion of intervention and 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Project HEART | Control: Project Growing Minds
Number analyzed (Participants) | 107 | 114
units on a scale | 3.62 (.47) | 3.51 (.46)
Statistical Analysis 1: Comparison: Project HEART vs Control: Project Growing Minds; Third, to assess the effectiveness of the HEART intervention from pretest to immediate posttest, we used linear regression analyses to compute adjusted means and mean differences between intervention and control groups. We included an indicator for school to adjust for clustering by school. For each outcome, the corresponding pretest measure was included as a covariate; Test type: Superiority — Before the onset of the study, we conducted a power calculation to determine the appropriate sample size. We designed the study to have 80% power at a .05 significance level to detect differences in primary outcomes, assuming an effect size of 0.5 and a correlation of 0.4 between assessments. Final enrollment (n= 222) exceeded our target sample size (n= 150); p = .32, Regression, Linear; beta = 0.05, Standard Error of Mean 0.05

3. Primary Outcome: 3-item Self-report of Sexual Communication Intentions Over Next 3 Months
Description: We assessed intentions to communicate about sex with items from the AIDS Risk Behavior Assessment. Three items captured the likelihood of communicating with a partner in the next 3 months about (1) sexual limits and boundaries, (2) STDs and pregnancy, and (3) condom use. Options ranged from 0% to 100% to indicate the likelihood of communicating with a partner. We averaged scores to create a composite (possible range 0-100); higher scores indicated greater likelihood of sexual communication (alpha = 0.84).
Time Frame: Immediate post-test at completion of intervention and 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Project HEART | Control: Project Growing Minds
Number analyzed (Participants) | 107 | 114
units on a scale | 87.0 (22.5) | 78.5 (27.9)
Statistical Analysis 1: Comparison: Project HEART vs Control: Project Growing Minds; We used linear regression analyses to compute adjusted means and mean differences between intervention and control groups. We included an indicator for school to adjust for clustering by school. For each outcome, the corresponding pretest measure was included as a covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < .001, Regression, Linear; beta = 8.31, Standard Error of Mean 2.71

ADVERSE EVENTS:
Groups:
- Project HEART: Interactive website with five modules to address safer sex motivation, knowledge, attitudes/norms, self-efficacy, and sexual communication skills. Program takes approximately 30-45 minutes to complete.
  Safer Sex: Interactive web-based intervention with five modules: motivation, knowledge, attitudes/norms, self-efficacy, and sexual communication skills.
  No adverse events.
- Control: Project Growing Minds: Attention-matched control website with five modules to address an introduction to mindsets, growth mindsets of intelligence, growth mindsets of self-control, growth mindsets of people, and an integrative summary. Program takes approximately 30-45 minutes to complete.
  Growth Mindsets: Interactive web-based intervention with five modules: mindsets introduction, growth mindsets of intelligence, growth mindsets of self-control, growth mindsets of people, and integrative summary.
  No adverse events.
Arm/Group | Project HEART | Control: Project Growing Minds
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/115
Other Adverse Events (participants affected / at risk) | 0/107 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No